CLINICAL TRIAL: NCT07278024
Title: To Investigate the Effect of Postbiotic Intervention on Vaginal Microbiota in Infertile Women
Brief Title: Postbiotic Intervention on Vaginal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Attending doctor, Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH25-CT1-18
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Infertile Women Undergoing IVF or ICSI
Keywords: vaginal microbiome; postbiotics; antimicrobial peptides; infertility; assisted reproductive technology; in vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postbiotics (Experimental)
  Interventions: Other: postbiotics

INTERVENTIONS:
Other: postbiotics — Participants will self-administer postbiotic intervention via intravaginal suppositories containing purified bacteriocin peptides . The intervention consists of one suppository administered intravaginally at bedtime, once daily for 8 consecutive weeks (56 days total). Each suppository contains a standardized concentration of bacteriocins extracted from Lactobacillus strains.

SUMMARY:
This study investigates the effects of postbiotic intervention on vaginal microbiota in infertile patients. Using a pre-post test design, we will enroll 15 women aged 30-45 years with at least two IVF failures. Participants will receive postbiotic intervention for 8 weeks. Vaginal secretion samples will be collected before and after treatment for 16S rRNA sequencing analysis to assess microbial composition, dominant species distribution, α-diversity index, and Lactobacillus content. Primary outcomes include changes in vaginal microbiota composition and diversity, alterations in Lactobacillus abundance, and pregnancy rates in subsequent IVF-FET cycles.

DETAILED DESCRIPTION:
Background The demand for infertility treatment is increasing, with approximately 10-15% of couples of reproductive age experiencing varying degrees of fertility issues. Vaginal microbiota dysbiosis may be a significant factor contributing to infertility, and a healthy vaginal microbiota environment plays a crucial role in embryo implantation. This study aims to investigate the effects of postbiotic intervention on the vaginal microbiota of infertile patients by analyzing the vaginal microbiota before and after bacteriocin treatment to evaluate its effectiveness in improving the vaginal microbial environment.

Objective This study aims to investigate changes in vaginal microbiota before and after the use of postbiotic intervention.

Methods This study employs a pre-post test design, planning to enroll 15 women aged 30-45 years diagnosed with infertility with at least two IVF treatment failure. All subjects must be free from severe gynecological diseases, not using antibiotics or probiotics, and without acute vaginal infection symptoms. The study period is 8 weeks. Before intervention, baseline data collection will include complete medical history and infertility treatment records. During the first visit, vaginal secretion samples will be collected for vaginal microbiota assessment through 16S rRNA sequencing analysis, simultaneously measuring Lactobacillus content and microbial diversity. Subjects will then use postbiotic intervention continuously for 8 weeks. After treatment, a second sampling will be conducted to re-analyze the vaginal microbiota. The primary outcome measures include changes in microbial composition before and after use, including dominant species distribution, α-diversity index, and changes in Lactobacillus content. All specimens will be collected, transported, and preserved following standard operating procedures to ensure testing quality. Research data will be analyzed using paired sample statistical methods to assess pre-post treatment differences, with significance level set at p<0.05.

Outcome

1. Compare differences in vaginal microbiota before and after using postbiotic intervention.
2. Compare differences in taxonomic abundance before and after using postbiotic intervention.
3. Check pregnancy rate of IVF-FET cycle after postbiotic intervention use

ELIGIBILITY:
Inclusion Criteria:

* (1) age 30-45 years;
* (2) body mass index 18-30 kg/m²;
* (3) history of ≥2 prior IVF treatment failures despite transfer of good-quality embryos;
* (4) planned FET cycle;
* (5) willingness to comply with the eight-week postbiotic intervention protocol

Exclusion Criteria:

* (1) active acute vaginal infection with symptomatic presentation;
* (2) antibiotic or probiotic use within the preceding three months;
* (3) congenital uterine anomalies including septate, bicornuate, or unicornuate uterus;
* (4) severe intrauterine adhesions (Asherman syndrome grade III-IV);
* (5) history of gynecologic malignancy;
* (6) known allergy or hypersensitivity to Lactobacillus-derived products;
* (7) current ongoing pregnancy

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Vaginal microbiome composition (genus level) | Baseline (Week 0) and post-intervention (Week 8)
  Changes in vaginal bacterial community structure assessed through 16S rRNA gene sequencing of vaginal secretion samples collected at baseline (Week 0) and post-intervention (Week 8)

SECONDARY OUTCOMES:
Taxonomic abundance (%) | Baseline (Week 0) and post-intervention (Week 8)
  Quantitative measurement of the relative proportions of bacterial taxa at different taxonomic levels (phylum, genus, and species) in vaginal samples before and after bacteriocin treatment. Results will report the percentage abundance of major bacterial groups.

OTHER OUTCOMES:
Pregnancy rate (%) | through study completion, an average of 8 months
  Visualization of fetal cardiac activity on transvaginal ultrasound at 6-7 weeks' gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar A, Green KM, Rawat M. A Comprehensive Overview of Postbiotics with a Special Focus on Discovery Techniques and Clinical Applications. Foods. 2024 Sep 17;13(18):2937. doi: 10.3390/foods13182937. PMID 39335866
- [Background] Vinderola G, Sanders ME, Salminen S. The Concept of Postbiotics. Foods. 2022 Apr 8;11(8):1077. doi: 10.3390/foods11081077. PMID 35454664
- [Background] Salminen S, Collado MC, Endo A, Hill C, Lebeer S, Quigley EMM, Sanders ME, Shamir R, Swann JR, Szajewska H, Vinderola G. The International Scientific Association of Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of postbiotics. Nat Rev Gastroenterol Hepatol. 2021 Sep;18(9):649-667. doi: 10.1038/s41575-021-00440-6. Epub 2021 May 4. PMID 33948025
- [Background] Moreno I, Garcia-Grau I, Perez-Villaroya D, Gonzalez-Monfort M, Bahceci M, Barrionuevo MJ, Taguchi S, Puente E, Dimattina M, Lim MW, Meneghini G, Aubuchon M, Leondires M, Izquierdo A, Perez-Olgiati M, Chavez A, Seethram K, Bau D, Gomez C, Valbuena D, Vilella F, Simon C. Endometrial microbiota composition is associated with reproductive outcome in infertile patients. Microbiome. 2022 Jan 4;10(1):1. doi: 10.1186/s40168-021-01184-w. PMID 34980280
- [Background] Zhao H, Wang C, Narsing Rao MP, Rafiq M, Luo G, Li S, Kang Y-Q. Effects of vaginal microbiota on in vitro fertilization outcomes in women with different infertility causes. Microbiol Spectr. 2025 Mar 4;13(3):e0125524. doi: 10.1128/spectrum.01255-24. Epub 2025 Jan 27. PMID 39868783
- [Background] Karaer A, Dogan B, Gunal S, Tuncay G, Arda Duz S, Unver T, Tecellioglu N. The vaginal microbiota composition of women undergoing assisted reproduction: a prospective cohort study. BJOG. 2021 Dec;128(13):2101-2109. doi: 10.1111/1471-0528.16782. Epub 2021 Jun 20. PMID 34053157
- [Background] Tian Q, Jin S, Zhang G, Liu Y, Liu J, Tang X, Li Y, Liu J, Liu Y, Wang Z. Assessing vaginal microbiome through Vaginal Microecology Evaluation System as a predictor for in vitro fertilization outcomes: a retrospective study. Front Endocrinol (Lausanne). 2024 Jul 9;15:1380187. doi: 10.3389/fendo.2024.1380187. eCollection 2024. PMID 39045277
- [Background] Su W, Gong C, Zhong H, Yang H, Chen Y, Wu X, Jin J, Xi H, Zhao J. Vaginal and endometrial microbiome dysbiosis associated with adverse embryo transfer outcomes. Reprod Biol Endocrinol. 2024 Aug 28;22(1):111. doi: 10.1186/s12958-024-01274-y. PMID 39198832
- [Background] Vainamo S, Saqib S, Kalliala I, Kervinen K, Luiro K, Niinimaki M, Halttunen-Nieminen M, Virtanen S, Nieminen P, Salonen A, Holster T. Longitudinal analysis of vaginal microbiota during IVF fresh embryo transfer and in early pregnancy. Microbiol Spectr. 2023 Dec 12;11(6):e0165023. doi: 10.1128/spectrum.01650-23. Epub 2023 Oct 26. PMID 37882794
- [Background] Onderdonk AB, Delaney ML, Fichorova RN. The Human Microbiome during Bacterial Vaginosis. Clin Microbiol Rev. 2016 Apr;29(2):223-38. doi: 10.1128/CMR.00075-15. PMID 26864580
- [Background] Gao X, Louwers YV, Laven JSE, Schoenmakers S. Clinical Relevance of Vaginal and Endometrial Microbiome Investigation in Women with Repeated Implantation Failure and Recurrent Pregnancy Loss. Int J Mol Sci. 2024 Jan 3;25(1):622. doi: 10.3390/ijms25010622. PMID 38203793
- [Background] Koedooder R, Singer M, Schoenmakers S, Savelkoul PHM, Morre SA, de Jonge JD, Poort L, Cuypers WJSS, Beckers NGM, Broekmans FJM, Cohlen BJ, den Hartog JE, Fleischer K, Lambalk CB, Smeenk JMJS, Budding AE, Laven JSE. The vaginal microbiome as a predictor for outcome of in vitro fertilization with or without intracytoplasmic sperm injection: a prospective study. Hum Reprod. 2019 Jun 4;34(6):1042-1054. doi: 10.1093/humrep/dez065. PMID 31119299
- [Background] Moreno I, Codoner FM, Vilella F, Valbuena D, Martinez-Blanch JF, Jimenez-Almazan J, Alonso R, Alama P, Remohi J, Pellicer A, Ramon D, Simon C. Evidence that the endometrial microbiota has an effect on implantation success or failure. Am J Obstet Gynecol. 2016 Dec;215(6):684-703. doi: 10.1016/j.ajog.2016.09.075. Epub 2016 Oct 4. PMID 27717732